CLINICAL TRIAL: NCT05799677
Title: The Effect of Reflexology in Patients With Viral Bronchiolitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Principal Investigator, Erez Nadir, MD, Principal Investigator, Hillel Yaffe Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0135-22-HYMC-IL
Record Dates: First submitted 2023-03-22; First posted 2023-04-05 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-04

CONDITIONS: Bronchiolitis; Chemical; Reflexology
Keywords: Bronchiolitis; Reflexology
MeSH Terms: conditions — Bronchiolitis | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Intervention Model Description: Comparing the extent of bronchiolitis between reflexology additive treatment to no reflexology treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reflexology (Experimental): Additive treatment with reflexology
  Interventions: Other: Reflexology
- Control (No Intervention): No treatment with reflexology

INTERVENTIONS:
Other: Reflexology — Additive reflexology treatment
  Arms: Reflexology

SUMMARY:
To test the influence of reflexology on bronchiolitis.

DETAILED DESCRIPTION:
Reflexology has been used in different respiratory tract infections on pulmonary function tests in patients with asthma, with some success. It has also been tested in newborns with respiratory distress syndrome, where it has decreased respiratory rate. Whole body massage was found to be helpful in newborns with opioid withdrawal syndrome. It has been shown to be a safe treatment and well tolerated even among very young infants.

Therefore, the investigators decided to evaluate effect of reflexology treatment in patients with viral bronchiolitis.

ELIGIBILITY:
Inclusion Criteria:

* All children admitted due to bronchiolitis

Exclusion Criteria:

* Children whose parents refused participation

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Hospitalization period | 1-14 days
  The time from admission to discharge (days)
Oxygen therapy period | 1-14 Days
  Number of days of oxygen treatment

CONTACTS AND LOCATIONS:
Overall Officials: Erez Nadir, MD, Principal Investigator — Hillel Yaffe Medical Center
Locations (1):
- Hillel Yaffe medical center, Hadera, Hadera, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fattah MA, Hamdy B. Pulmonary functions of children with asthma improve following massage therapy. J Altern Complement Med. 2011 Nov;17(11):1065-8. doi: 10.1089/acm.2010.0758. PMID 22087616
- [Background] Miralizadeh A, Peyman A, Jamali Soltani N, Ashktorab T. Comparison of the Effect of Foot and Palm Reflexology Massage on Respiratory Distress Syndrome in Premature Infants under Noninvasive Ventilation. Complement Med Res. 2022;29(2):100-108. doi: 10.1159/000517982. Epub 2021 Oct 29. PMID 34818220
- [Background] Rana D, Garde K, Elabiad MT, Pourcyrous M. Whole body massage for newborns: A report on non-invasive methodology for neonatal opioid withdrawal syndrome. J Neonatal Perinatal Med. 2022;15(3):559-565. doi: 10.3233/NPM-220989. PMID 35599503
- [Background] Jones LM, Regan C, Wolf K, Bryant J, Rakowsky A, Pe M, Snyder DA. Effect of osteopathic manipulative treatment on pulmonary function testing in children with asthma. J Osteopath Med. 2021 May 7;121(6):589-596. doi: 10.1515/jom-2020-0040. PMID 33962511
- [Background] Roque i Figuls M, Gine-Garriga M, Granados Rugeles C, Perrotta C, Vilaro J. Chest physiotherapy for acute bronchiolitis in paediatric patients between 0 and 24 months old. Cochrane Database Syst Rev. 2016 Feb 1;2(2):CD004873. doi: 10.1002/14651858.CD004873.pub5. PMID 26833493
- [Background] Wang EE, Milner RA, Navas L, Maj H. Observer agreement for respiratory signs and oximetry in infants hospitalized with lower respiratory infections. Am Rev Respir Dis. 1992 Jan;145(1):106-9. doi: 10.1164/ajrccm/145.1.106. PMID 1731571